CLINICAL TRIAL: NCT03977259
Title: Targeting Human Milk Fortification to Improve Preterm Infant Growth and Brain Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mandy Brown Belfort, MD MPH, Attending physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2019P000893
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Preterm Birth; Breast Milk Expression; Nutrition Disorder, Infant; Brain Development Abnormality; Neurodevelopmental Disorders
MeSH Terms: conditions — Premature Birth; Breast Milk Expression; Infant Nutrition Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parents, clinical, and research staff apart from the study milk technician will be unaware of the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard fortification (No Intervention): Standard of care fortification with multicomponent human milk fortifier (24 kcal/oz) and liquid protein (0.27 g/dL); additional protein and/or calories added only for growth faltering.
- Individually targeted fortification (Experimental): Standard of care fortification plus extra protein and/or calories to ensure that "base" milk has protein 1 g/dL and calories 67/dL.
  Interventions: Other: Individually targeted fortification

INTERVENTIONS:
Other: Individually targeted fortification — Abbott liquid protein and/or medium chain triglyceride are added routinely to ensure that the "base" milk has protein 1 g/dL and calories 67/dL.
  Arms: Individually targeted fortification

SUMMARY:
This study is a randomized trial comparing 2 methods of human milk fortification for preterm infants in the neonatal intensive care unit (NICU). All participating infants will receive a human milk diet comprising maternal and/or donor milk plus multi-component and modular fortifiers. In one group (control), the milk will be fortified according to routine standard of care. In the other group (intervention), the fortification will be individually targeted based on the results of point-of-care human milk analysis. Outcomes include physical growth in the NICU and after discharge, brain structure by magnetic resonance imaging at term equivalent age, and neurodevelopment at 2 years.

DETAILED DESCRIPTION:
Human milk is the recommended diet for preterm infants and it requires fortification to meet their high nutrient requirements. This study addresses a gap in knowledge about the optimal strategy for human milk fortification in the neonatal intensive care unit (NICU).

Infants will be recruited from a single site (Brigham and Women's Hospital, Boston MA). Eligible infants are NICU inpatients born <31 weeks' gestation and enrolled within 21 days of birth, whose mothers are providing breast milk. Exclusion criteria include major congenital anomalies, severe fetal growth restriction (weight <3rd percentile), clinically significant gastrointestinal pathology, triplets or higher order multiples, and expected death or transfer. Infants who require fluid restriction <140 mL/kg/day will also be excluded.

The study period begins when infants have reached full volume (150-160 mL/kg/day) human milk feedings fortified to 24 kcal per ounce. Participants will be randomized to one of two diet groups; twins will be randomized separately. The study diet will continue until 36 weeks' postmenstrual age or hospital discharge, whichever comes first.

Available maternal milk will be pooled with donor milk (if needed) to reach the total daily fluid volume; this "base" milk will be analyzed with a point-of-care human milk analyzer (Miris, AB). All infants will receive at minimum the standard human milk fortification (multicomponent fortifier to 24 kcal/oz plus liquid protein 0.27 g/dL). In one group (control), we will follow the standard of care for milk fortification, only adding more protein and/or energy if weight gain is lagging. In the other group (intervention), we will individually target fortification with additional protein and/or energy so that the "base" milk always contains protein 1 g/dL and energy 67 kcal/dL.

Outcome measures will include physical growth during the diet intervention period, including gain in weight, length, and head circumference and body composition with air displacement plethysmography at the end of the diet intervention. At term equivalent age, participants will undergo brain magnetic resonance imaging. At 2 years corrected age, outcomes include standard and novel neurodevelopmental tests including the Bayley-III and tests of emerging executive function; and physical size.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient in Brigham and Women's Hospital NICU
* Gestational age 24 0/7 to 30 6/7 weeks
* Chronologic age <21 days
* Mother providing breast milk

Exclusion Criteria:

* Major congenital anomaly
* Severe fetal growth restriction (birth weight <3rd percentile by Olsen reference)
* Necrotizing enterocolitis, intestinal perforation, other major gastrointestinal pathology
* Triplets or higher order multiples
* Plan for redirection of care and/or anticipated death
* Clinically significant renal or hepatic dysfunction
* Inborn error of metabolism
* Fluid restriction <140 mL/kg/day for 3 or more days
* Grade 3 or 4 intraventricular hemorrhage detected prior to enrollment
* Anticipated transfer <36 weeks' postmenstrual age
* Parents do not consent to use of pasteurized donor human milk
* Infant in non-parental custody

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight | at study endpoint (36 weeks' postmenstrual age or discharge)
  Weight z-score
Length | at study endpoint (36 weeks' postmenstrual age or discharge)
  Length z-score
Fat free mass | at study endpoint (36 weeks' postmenstrual age or discharge)
  Fat free mass estimated with air displacement plethysmography (z-score)
Total brain volume | at term equivalent age (38 to 41 weeks' postmenstrual age)
  Total brain volume by MRI
Cerebellar volume | at term equivalent age (38 to 41 weeks' postmenstrual age)
  Cerebellar volume by MRI
Bayley-III cognitive score | at 2 years' corrected age
  Scaled composite score (continuous), higher score indicates better performance, range of possible scores 55-145
Bayley-III motor score | at 2 years' corrected age
  Scaled composite score (continuous), higher score indicates better performance, range of possible scores 46-154

SECONDARY OUTCOMES:
Fat mass | at study endpoint (36 weeks' postmenstrual age or discharge)
  Fat mass estimated with air displacement plethysmography (z-score)
Weight | at 2 years' corrected age
  Weight z-score
Height | at 2 years' corrected age
  Height z-score
Low Bayley-III cognitive score | At 2 years' corrected age
  Scaled composite score <85 (>1 standard deviation below the normative mean)
Low Bayley-III motor score | At 2 years' corrected age
  Scaled composite score <85 (>1 standard deviation below the normative mean)
Bayley-III language score | At 2 years' corrected age
  Scaled composite score (continuous), higher score indicates better performance, range of possible scores 46-154
Bayley-III language score | At 2 years' corrected age
  Scaled composite score <85 (>1 standard deviation below the normative mean)
Spacial working memory | at 2 years' corrected age
  Spin the Pots task (number of trials, search time)
Behavioral inhibition | at 2 years' corrected age
  Mommies and Babies task (number of trials, errors)
Executive function | at 2 years' corrected age
  Behavioral Rating Inventory of Executive Function - Preschool Version, higher scores indicate more problems
Behavioral difficulties | at 2 years' corrected age
  Infant-Toddler Symptom Checklist - Long Version, higher scores indicate more problems

CONTACTS AND LOCATIONS:
Overall Officials: Mandy B Belfort, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No current plans to share individual patient data. Future data sharing would involve de-identified data only and would require a data use agreement in accordance with hospital policy.

REFERENCES:
- [Derived] Belfort MB, Woodward LJ, Cherkerzian S, Pepin H, Ellard D, Steele T, Fusch C, Grant PE, Inder TE. Targeting human milk fortification to improve very preterm infant growth and brain development: study protocol for Nourish, a single-center randomized, controlled clinical trial. BMC Pediatr. 2021 Apr 9;21(1):167. doi: 10.1186/s12887-021-02635-x. PMID 33836708